CLINICAL TRIAL: NCT04177836
Title: Mindfulness and Romantic Relationship Quality
Acronym: MINDv2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Lisa Jaremka, Principal Investigator, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R21AT010515-01 (NIH)
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: The Focus of the Study is Romantic Relationship Quality
Keywords: Romantic relationship quality; Mindfulness

STUDY DESIGN:
Intervention Model Description: There are 2 arms to this intervention - mindfulness and active control.
Who Masked: Participant
Masking Description: The participant and the people interacting with participants will be blind to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIndfulness (Experimental): This arm was developed to increase attention towards and acceptance of current experiences.
  Interventions: Behavioral: Mindfulness intervention
- Active Control (Active Comparator): This arm is a relaxation-based active treatment comparison intervention, developed to parallel the structure of the mindfulness intervention without the attention towards or acceptance of present experiences.
  Interventions: Behavioral: Mindfulness intervention

INTERVENTIONS:
Behavioral: Mindfulness intervention — Participants will either complete a mindfulness intervention or active control for 2 weeks on their smartphone

SUMMARY:
The overarching aim of this proposal is to experimentally test whether a mindfulness intervention improves relationship quality. Romantic couples from the community will be randomly assigned to one of two arms: mindfulness vs. active control. Both interventions will be completed on a smart-phone for 14 days using identical intervention activities as our existing published research. After the 14-day period, couples will attend a lab visit and provide relationship quality data.

DETAILED DESCRIPTION:
Romantic couples from the community will be randomly assigned to one of two arms: mindfulness vs. active control. Thus, both partners will either complete the mindfulness intervention (developed to increase attention towards and acceptance of current experiences) or a relaxation-based active treatment comparison intervention (developed to parallel the structure of the mindfulness intervention without the attention towards or acceptance of present experiences). Both interventions will be completed on a smart-phone for 14 days using identical intervention activities as our existing published research, which demonstrated that the mindfulness intervention reduced stress reactivity and improved daily well-being. After the 14-day period, couples will attend a lab visit and provide multi-method relationship quality data.

ELIGIBILITY:
Inclusion Criteria:

* Couples living together for at least 2 years
* Both partners must be fluent in English
* Both partners cannot already engage in regular systematic mind-body practice (>2 times per week).
* Both partners must have daily access to an internet-enabled smartphone to complete the intervention

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Romantic Relationship Quality | Before and after the 2 week intervention
  Assessed with well validated sel-report questionnaire, the Couples Satisfaction Index

SECONDARY OUTCOMES:
Changes in Sleep quality | Before and after the 2 week intervention
  Assessed with well validated measure, the PROMIS sleep disturbance questionnaire
Changes in Depressive symptoms | Before and after the 2 week intervention
  Assessed with well validated measure, the PROMIS depressive symptoms questionnire
Changes in Blood pressure | Before and after the 2 week intervention
  Assessed with well validated measure, physiological assessment via a blood pressure machine
Changes in Life satisfaction | Before and after the 2 week intervention
  Assessed with well validated measure, the Life Satisfaction Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
We will not share IPD.